CLINICAL TRIAL: NCT01576224
Title: Early Mobilization After Volar Plate Osteosynthesis of Distal Radius Fractures. A Prospective Randomized Study.
Brief Title: Early Mobilization After Volar Plate Osteosynthesis of Distal Radius Fractures
Acronym: E-MOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Region Sjællands sundhedsvidenskabelige Forskningsfond (Unknown)
Responsible Party: Principal Investigator, Thomas Juul Sørensen, Principal Investigator, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SJ-275
Record Dates: First submitted 2012-04-09; First posted 2012-04-12 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Distal Radius Fracture
Keywords: Volar locking plate osteosynthesis; Early mobilization; DASH
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate mobilization (Experimental): Patients start exercises immediately after osteosynthesis.
  Interventions: Device: Removable splint "omni med", Fischer Medical Aps, DK-2800 Lyngby, Denmark
- Later mobilization (Active Comparator): Patients are allowed exercises after 14 days.
  Interventions: Device: Removable splint "omni med", Fischer Medical Aps, DK-2800 Lyngby, Denmark

INTERVENTIONS:
Device: Removable splint "omni med", Fischer Medical Aps, DK-2800 Lyngby, Denmark — To be removed during training exercises three to five times a day

SUMMARY:
The aim of this study is to investigate the post operational mobilization after volar locking plate osteosynthesis of distal radius fractures. One group is admitted training exercises just after the fracture treatment, one group after 14 days immobilization in a cast.

The primary hypothesis is, that immediate training leads to earlier and faster recovery.

Our second hypothesis is, that immediate training does not lead to increased risk of fracture displacement.

DETAILED DESCRIPTION:
Patients were followed for one year with controls after one, three, six and twelve months. Occupational therapists blinded for the intervention examined the patients at all times. ROM, strength and DASH score was performed.

ELIGIBILITY:
Inclusion Criteria:

* Over 50 years of age
* Distal radius fracture suitable for volar locking plate osteosynthesis
* Inhabitants in Region Sjaelland

Exclusion Criteria:

* Dementia
* Abuse of drugs, medication or alcohol
* Open fractures
* Multitrauma or other injures on same extremity
* Earlier wrist fracture
* Delay of osteosynthesis of more than 14 days

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Disability of arm, shoulder and hand score (DASH) | After 4 weeks
Disability of arm, shoulder and hand score (DASH) | After 3 months
Disability of arm, shoulder and hand score (DASH) | After 6 months
Disability of arm, shoulder and hand score (DASH) | After 12 months

SECONDARY OUTCOMES:
Range of motion | After 4 weeks
Range of motion | After 3 months
Range of motion | After 6 months
Range of motion | After 12 months
Grip strength | After 4 weeks
Grip strength | After 3 months
Grip strength | After 6 months
Grip strength | After 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Sørensen, Consultant, Principal Investigator — Køge Sygehus, Denmark
Locations (1):
- Køge Sygehus, Køge, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No